CLINICAL TRIAL: NCT05873712
Title: A Phase II Study Evaluating the Safety and Efficacy of the Combination of Zanubrutinib Plus Lisocabtagene Maraleucel for Richter's Syndrome
Brief Title: Zanubrutinib and Lisocabtagene Maraleucel for the Treatment of Richter's Syndrome
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Aseel Alsouqi (Other)
Collaborators: BeOne Medicines (Industry)
Responsible Party: Sponsor-Investigator, Aseel Alsouqi, Principal Investigator, Ohio State University Comprehensive Cancer Center
Organization: Ohio State University Comprehensive Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSU-22157; NCI-2023-03669 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2023-05-15; First posted 2023-05-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Recurrent Transformed Chronic Lymphocytic Leukemia; Refractory Transformed Chronic Lymphocytic Leukemia; Transformed Chronic Lymphocytic Leukemia to Diffuse Large B-Cell Lymphoma; Recurrent Transformed B-Cell Non-Hodgkin Lymphoma; Recurrent Transformed Non-Hodgkin Lymphoma; Refractory Transformed Non-Hodgkin Lymphoma; Refractory Transformed B-cell Non-Hodgkin Lymphoma; Refractory Transformed
Keywords: Richter's Transformation; Richter's Syndrome
MeSH Terms: interventions — Specimen Handling; Biopsy; Cyclophosphamide; fludarabine; Leukapheresis; Sentinel Lymph Node Biopsy; Magnetic Resonance Spectroscopy; zanubrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (zanubrutinib, liso-cel) (Experimental): Patients receive zanubrutinib PO, undergo leukaphereis, and receive fludarabine IV, cyclophosphamide IV, and liso-cel IV on study. Patients also undergo BM biopsy and lymph node biopsy at screening and follow up, and undergo collection of blood samples and CT, PET/CT, and/or MRI throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Biopsy; Procedure: Computed Tomography; Drug: Cyclophosphamide; Drug: Fludarabine; Procedure: Leukapheresis; Biological: Lisocabtagene Maraleucel; Procedure: Lymph Node Biopsy; Procedure: Positron Emission Tomography; Drug: Zanubrutinib

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of blood samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Marrow Biopsy — Undergo BM biopsy
  Other Names: Biopsy of Bone Marrow; Biopsy, Bone Marrow
Procedure: Computed Tomography — Undergo CT and/or PET/CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; CT; CT Scan; tomography
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
Drug: Fludarabine — Given IV
  Other Names: Fluradosa
Procedure: Leukapheresis — Given IV
  Other Names: Leukocytopheresis; Therapeutic Leukopheresis
Biological: Lisocabtagene Maraleucel — Given IV
  Other Names: Anti-CD19-CAR Genetically Engineered Autologous T Lymphocytes JCAR017; Anti-CD19-CAR Genetically Engineered Autologous T-lymphocytes JCAR017; Autologous Anti-CD19-EGFRt-4-1BB-zeta-modified CAR CD8+ and CD4+ T-lymphocytes JCAR017; Breyanzi; JCAR 017; JCAR017
Procedure: Lymph Node Biopsy — Undergo lymph node biopsy
  Other Names: Biopsy of Lymph Node
Procedure: Positron Emission Tomography — Undergo PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging; PT
Drug: Zanubrutinib — Given PO
  Other Names: BGB-3111; Brukinsa; BTK-InhB

SUMMARY:
This phase II trial tests how well zanubrutinib and lisocabtagene maraleucel (liso-cel) work together in treating patients with Richter's syndrome. Richter's syndrome occurs when chronic lymphocytic leukemia and/or small lymphocytic leukemia transforms into an aggressive lymphoma, which is a cancer of the lymph nodes. Zanubrutinib is a class of medication called a kinase inhibitor. These drugs work by preventing the action of abnormal proteins that tell cancer cells to multiply, which helps stop the spread of cancer. Liso-cel is a type of treatment known as chimeric antigen receptor (CAR) T cell therapy. CAR T-cell therapy is a type of treatment in which a patient's T cells (a type of immune system cell) are changed in the laboratory so they will attack cancer cells. T cells are taken from a patient's blood. Then the gene for a special receptor that binds to a certain protein on the patient's cancer cells is added to the T cells in the laboratory. The special receptor is called a chimeric antigen receptor (CAR). Large numbers of the CAR T cells are grown in the laboratory and given to the patient by infusion for treatment of certain cancers. Giving zanubrutinib and liso-cell together may kill more cancer cells in patients with Richter's syndrome.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the efficacy of the combination of zanubrutinib and lisocabtagene maraleucel (liso-cel) for the treatment of Richter's syndrome (RS).

SECONDARY OBJECTIVES:

I. To describe the safety profile of the combination of zanubrutinib and liso-cel for RS.

II. To evaluate duration of the efficacy of the combination of zanubrutinib and liso-cel for RS

CORRELATIVE OBJECTIVES:

I. Describe T-cell subsets before and after zanubrutinib initiation, as well as post liso-cel infusion.

II. To describe the persistence of liso-cel. III. To describe the tumor microenvironment post liso-cel infusion at relapse. IV. Investigate the correlation between inflammatory cytokines and measures of inflammation and outcomes and rates of adverse events including cytokine release syndrome (CRS).

V. Investigate chronic lymphocytic leukemia (CLL) persistence post treatment.

OUTLINE:

Patients receive zanubrutinib orally (PO), undergo leukaphereis, and receive fludarabine intravenously (IV), cyclophosphamide IV, and liso-cel IV on study. Patients also undergo bone marrow (BM) biopsy and lymph node biopsy at screening and follow up, and undergo collection of blood samples and computed tomography (CT), positron emission tomography (PET)/CT, and/or magnetic resonance imaging (MRI) throughout the trial.

After study completion, patients are followed for 24 months, and then every 6 months until disease progression or death.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of RS - occurrence of diffuse large B-cell lymphoma (DLBCL) in patients with antecedent or concurrent CLL/SLL (CLL/SLL diagnosis per IWCLL 2018 criteria).
* Must have relapsed/refractory disease as defined by one of the following:

  * Participants must have undergone >= 1 prior systemic therapeutic regimen administered for >= 1 cycle for either CLL or RS, and have had either documented disease progression to the most recent treatment regimen, or refractory disease. OR
  * Developed RS while receiving treatment for CLL
* Age >= 18 years
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Total bilirubin =< 2.0 times the institutional upper limit of normal (unless documented Gilbert's syndrome)
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT]) =< 2.5 x institutional upper limit of normal
* Alanine aminotransferase (ALT) (serum glutamic-pyruvic transaminase [SGPT]) =< 2.5 x institutional upper limit of normal
* Creatinine clearance >= 30 mL/min

  * Using 24-hour creatinine clearance or standard Cockcroft-Gault equation
* Absolute lymphocyte count > 100/uL at screening
* Left ventricular ejection fraction >= 40% by multigated acquisition (MUGA) or echocardiogram (ECHO)
* Adequate bone marrow independent of growth factor support or infusion support at screening unless evidence shows that the cytopenia(s) is due to marrow involvement by CLL/small lymphocytic lymphoma (SLL). If cytopenias are due to disease in the bone marrow any degree of anemia or thrombocytopenia are allowed, absolute neutrophil count (ANC) must be >= 500
* Absolute neutrophil count (ANC) >= 1000/mm^3 (independent of growth factor support or infusion support at screening unless evidence shows that the cytopenia[s] is due to marrow involvement by CLL/SLL). If cytopenias are due to disease in the bone marrow any degree of anemia or thrombocytopenia are allowed, ANC must be >= 500
* Platelets >= 30,000/mm^3 (independent of growth factor support or infusion support at screening unless evidence shows that the cytopenia[s] is due to marrow involvement by CLL/SLL). If cytopenias are due to disease in the bone marrow any degree of anemia or thrombocytopenia are allowed
* Hemoglobin >= 7 g/dL (independent of growth factor support or infusion support at screening unless evidence shows that the cytopenia[s] is due to marrow involvement by CLL/SLL). If cytopenias are due to disease in the bone marrow any degree of anemia or thrombocytopenia are allowed
* Radiographically measurable lymphadenopathy (or measurable extra-nodal disease) per Lugano criteria
* Must meet all institutional standards for receiving CAR T-cell therapy
* Subjects (or legal guardians) must have the ability to understand and the willingness to sign a written informed consent document
* For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use a contraceptive method with a failure rate of < 1% per year, initiated prior to first dose of study drug, during the treatment period and for at least 1 year after the CAR-T cell infusion or 1 month after last dose of zanubrutinib, whichever is longer.

  * A woman is considered to be of childbearing potential if she is postmenarcheal, has not reached a postmenopausal state (< 12 continuous months of amenorrhea with no identified cause other than menopause), and has not undergone surgical sterilization (removal of ovaries and/or uterus). Examples of contraceptive methods with a failure rate of < 1% per year include bilateral tubal ligation, male sterilization, hormonal contraceptives that inhibit ovulation, hormone-releasing intrauterine devices, and copper intrauterine devices
* For men: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures, and agreement to refrain from donating sperm, as defined below:

  * With female partners of childbearing potential, men must remain abstinent or use a condom plus an additional contraceptive method that together result in a failure rate of < 1% per year during the treatment period and for at least 1 year after the anti-CD19 CAR-T cell infusion or 1 month after last dose of zanubrutinib, whichever is longer. Men should avoid fathering a child and refrain from donating sperm during this same period.
  * With pregnant female partners, men must remain abstinent or use a condom during the treatment period and for at least 1 year after the human anti- CD19 CAR-T cell infusion or 1 month post last dose of zanubrutinib, whichever is longer, to avoid potential embryonal or fetal exposure. The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not acceptable methods of contraception

Exclusion Criteria:

* A history of treatment including any of the following: prior CD19 directed therapy, treatment with alemtuzumab within 6 months before enrollment, prior allogeneic hematopoietic stem cell transplant (SCT) or donor lymphocyte infusion (DLI) within 2 months prior to enrollment
* Prior allogeneic stem cell transplant with active graft-versus-host disease (GVHD), or requiring immunosuppressive drugs for treatment of GVHD, or have taken calcineurin inhibitors within 4 weeks prior to consent
* Inadequate recovery from adverse events related to prior therapy to grade =< 1 (excluding grade 2 alopecia, neuropathy, and hypertension)
* Is unable to swallow oral medication, or has significant gastrointestinal disease that would limit absorption of oral medication
* Active bleeding or history of bleeding diathesis (e.g., hemophilia or von Willebrand disease)
* Uncontrolled autoimmune hemolytic anemia (AIHA) or idiopathic thrombocytopenic purpura (ITP)
* Presence of a gastrointestinal ulcer diagnosed by endoscopy within 3 months before screening
* Clinically significant cardiovascular disease such as symptomatic arrhythmias, congestive heart failure, or myocardial infarction within 6 months of screening, or any class 3 or 4 cardiac disease as defined by the New York Heart Association Functional Classification. Note: Subjects with controlled atrial fibrillation/flutter can enroll on study
* Requires or receiving anticoagulation with warfarin or equivalent vitamin K antagonists
* Prothrombin time (PT)/international normalized ratio (INR) or activated partial thromboplastin time (PTT) (in the absence of lupus anticoagulant) > 2 x upper limit normal (ULN)
* Treatment with a moderate or strong CYP3A inhibitor or inducer within 7 days prior to first dose of zanubrutinib
* Patients may not have an active intercurrent disease or concurrent malignancy that is expected to limit survival to < 5 years
* Human immunodeficiency virus (HIV) seropositivity at screening
* Subjects with uncontrolled intercurrent illness including, but not limited to ongoing or active infection, unstable angina pectoris, pulmonary abnormalities or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant or breastfeeding women are excluded from this study because CAR-T cell therapy may be associated with the potential for teratogenic or abortifacient effects. Women of childbearing potential must have a negative serum pregnancy test. Because there is an unknown, but potential risk for adverse events in nursing infants secondary to treatment of the mother with CAR-T cells, breastfeeding should be discontinued. These potential risks may also apply to other agents used in this study
* Evidence of myelodysplasia or cytogenetic abnormality indicative of myelodysplasia on any bone marrow biopsy prior to initiation of therapy
* Serologic status reflecting active hepatitis B or C infection at screening. Patients that are positive for hepatitis B core antibody, hepatitis B surface antigen (HBsAg), or hepatitis C antibody must have a negative polymerase chain reaction (PCR) at screening. PCR positive patients will be excluded
* History of autoimmune disease (i.e. rheumatoid arthritis, systemic lupus erythematosus) with requirement of immunosuppressive medication within 6 months
* Chronic use of corticosteroids >= 20mg prednisone equivalent PO daily
* Live vaccines given in 28 days prior to lymphodepleting chemotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-07-28 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall response rate | At 90 days after lisocabtagene maraleucel (liso-cel) infusion
  Overall response rate (ORR) will be defined as the proportion of patients achieving a complete or partial response divided by the number of efficacy-evaluable patients according to the Revised Response Criteria for Malignant Lymphoma. Response will be assessed using Lugano criteria 2014. ORR will be reported with two-sided 95% and 80% binomial exact confidence intervals.

SECONDARY OUTCOMES:
Incidence of adverse events | Up to 2 years
  Adverse event data will be collected on all patients who receive at least one dose of study drug(s). Non-hematologic adverse events (AEs) will be graded according to Common Terminology Criteria for Adverse Events version 5.0. Hematologic AEs will be graded according to chronic lymphocytic leukemia-specific criteria described in the International Workshop on Chronic Lymphocytic Leukemia 2018 guidelines.
Progression free survival | Time from liso-cel infusion until documented disease progression, or death from any cause, whichever occurs first, assessed up to 2 years
  Will be estimated using Kaplan-Meier methodology. Median estimates and estimates at clinically meaningful time points will be reported with 95% confidence intervals.
Overall survival | Time from liso-cel infusion until death from any cause, assessed up to 2 years
  Will be estimated using Kaplan-Meier methodology. Median estimates and estimates at clinically meaningful time points will be reported with 95% confidence intervals.
Duration of response | Time from the first tumor assessment that supports response to the time of confirmed disease progression or death due to any cause, whichever occurs first, assessed up to 2 years
  Will be estimated using Kaplan-Meier methodology. Median estimates and estimates at clinically meaningful time points will be reported with 95% confidence intervals.
Time to next treatment (TTNT) | Time from liso-cel infusion until next treatment is initiated, assessed up to 2 years
  Will be estimated using Kaplan-Meier methodology. TTNT will be estimated using the cumulative incidence competing risk method. Median TTNT and TTNT at clinically meaningful time points will be estimated and reported with 95% cumulative incidences.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer A Woyach, MD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (3):
- United States (3):
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Huntsman Cancer Institute, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu